CLINICAL TRIAL: NCT07353060
Title: Prognostic Profile of Dupuytren's Disease: a Cohort Study
Brief Title: Prognostic Profile of Dupuytren's Disease: a Cohort Study (PRODUCT)
Acronym: PRODUCT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ramsay Générale de Santé (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2024-A00473-44
Record Dates: First submitted 2026-01-13; First posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Dupuytren's Disease
MeSH Terms: conditions — Dupuytren Contracture | interventions — Surveys and Questionnaires; Restraint, Physical

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patient with Dupuytren's disease (Experimental): Treatment by percutaneous needle aponeurotomy
  Interventions: Other: Questionnaires; Other: Clinical examination

INTERVENTIONS:
Other: Questionnaires — The functional assessment of patients will be carried out using the Quick DASH, URAM and Southampton scores.
Other: Clinical examination — A clinical examination of the patient with assessment of the morphological impact by quantifying the deformity of the fingers in flexion using angular measurement and the Tubiana score

SUMMARY:
Dupuytren's disease is characterized by retractile fibrosis of the superficial palmar aponeurosis, which can lead to irreversible flexion contractures of the fingers and lasting functional impairment. Widespread throughout the world, it has a particularly high prevalence in northern European countries. This has been estimated at between 3.5% and 11% in England and Denmark. This prevalence is expected to increase over time due to the aging population. Risk factors for the disease include age, male sex, heredity, diabetes, smoking, and alcohol consumption. The resulting disability is not spontaneously reversible. It affects various aspects of daily life, most notably personal care, nutrition, and social interaction.

Treatment for Dupuytren's disease, whether medical or surgical, remains symptomatic to date and does not preclude the possibility of recurrence. In France, it is based on percutaneous needle aponeurotomy and surgical aponeurectomy. Its objectives are to reduce the flexion contracture of the fingers and the functional disability caused by the disease. Enzymatic aponeurosis with collagenase is also possible, but it is less well tolerated than percutaneous needle aponeurotomy. It is more expensive and not covered by health insurance.

The widespread adoption of a medical-surgical strategy that positions percutaneous needle aponeurotomy as the first-line treatment could improve the acceptability of Dupuytren's disease treatment and significantly reduce its cost to healthcare systems. However, the impact of this strategy depends on the extent to which second-line surgery is required. This use has been little studied. The proportion of patients requiring surgical treatment after percutaneous needle aponeurotomy is estimated to be 10 to 18%. These data are based on small sample sizes observed over varying follow-up periods. They need to be verified in large populations using a prospective study. Moreover, the factors associated with the need for surgery after percutaneous needle ablation for Dupuytren's disease are currently poorly understood. Understanding these factors would be beneficial for optimizing medical and surgical management. It could allow for better tailoring of treatment options to the patient's individual profile.

DETAILED DESCRIPTION:
Percutaneous needle aponeurotomy for Dupuytren's disease was developed by Jean-Luc Lermusiaux in 1972, in the Rheumatology Department of Lariboisière Hospital in Paris. Its efficacy, tolerability, simplicity, and low cost make it a standard treatment. For many, provided they are informed about the existence of this technique and master it, it is the first-line treatment for Dupuytren's disease. Within the framework of a graduated medical-surgical strategy, and in our practice, surgery for Dupuytren's disease therefore appears as a second-line treatment indicated in cases of failure after percutaneous treatment. This positioning is, however, not universally accepted. Surgery remains the most common treatment for Dupuytren's disease today.

The main objective of the study is to describe the proportion of patients requiring surgery within 3 years of treatment by percutaneous needle aponeurotomy for Dupuytren's disease

ELIGIBILITY:
Inclusion Criteria:

* Patient, male or female, over 18 years of age
* Patient with Dupuytren's disease confirmed by clinical examination: nodule or cord arising from the superficial palmar aponeurosis, visible or palpable
* Aponeurotic cord causing an MCP or PIP joint flexion contracture of at least 20°
* Indication for percutaneous needle ablation (flexion contracture of at least 20°, functionally impaired according to the patient)
* Acceptance of percutaneous needle ablation by the patient
* Patient affiliated with or covered by a social security scheme
* Patient having been informed and having signed a free and informed written consent
* Negative urine pregnancy test for women of childbearing age

Exclusion Criteria:

* Minor patient,
* Patient with another condition, infection, or wound of the hand,
* Patient participating in another clinical trial,
* Protected patient: adult under guardianship, curatorship, or other legal protection, deprived of liberty by judicial or administrative decision,
* Person unable to express their consent,
* Pregnant, breastfeeding, or parturient woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 305 (Estimated)
Dates: Start 2026-02-04 (Estimated); Primary Completion 2030-12-04 (Estimated); Study Completion 2031-02-04 (Estimated)

PRIMARY OUTCOMES:
Use of surgery (yes/no) | 3 years
  Use of surgery within 3 years following treatment by percutaneous needle aponeurotomy for Dupuytren's disease. the result is yes or not.

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Lariboisière, Paris, France